CLINICAL TRIAL: NCT03919279
Title: Transcutaneous Auricular Vagus Nerve Stimulation in Erosive Hand Osteoarthritis
Brief Title: Treatment of Erosive Digital Osteoarthritis by Transcutaneous Auricular Nerve Stimulation
Acronym: ADEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP190156
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Erosive Osteo-Arthritis; Hand Osteoarthritis
Keywords: Erosive hand osteoarthritis; pain; inflammation; vagus nerve stimulation
MeSH Terms: conditions — Pain; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- active arm with active tVNS for 1 month (Experimental)
  Interventions: Device: active tVNS

INTERVENTIONS:
Device: active tVNS — tVNS using TENS device from Schwa-Medico (TENSeco2) + auricular electrode applied on the left ear (Schwa-Medico) + conductive gel class I; 25 Hz stimulation 1 hour daily for 1 month

SUMMARY:
Erosive hand osteoarthritis (EHOA) is a subtype of had osteoarthritis characterized by inflammation and pain, with subsequent burden. Few symptomatic treatments are available in EHOA, while this population with EHOA has frequently comorbidities.

Stimulation of the vagus nerve (VN), belonging to parasympathetic system, dampens pro-inflammatory cytokines production by splenic macrophages, through to the binding of acetylcholine neurotransmitter to α7nicotinic receptor on macrophages: this is the cholinergic anti-inflammatory pathway (CAP). Beyond its anti-inflammatory effects, VNS is analgesic in chronic pain disorders (headache, fibromyalgia). Beside implantable devices, VNS may be performed using transcutaneous stimulation of the ascendant auricular branch of the VN (tVNS) at the left ear localized on the cymba conchae tVNS is well-tolerated therapy avoiding invasive neurosurgery.

The investigator do the hypothesis that auricular tVNS using a transcutaneous electrical nerve stimulation (TENS) device could be a novel, simple and well-tolerated analgesic and anti-inflammatory treatment of symptomatic EHOA.

DETAILED DESCRIPTION:
In symptomatic and inflammatory EHOA patients, we will apply tNVNS using device from Schwa-Medico (TENSeco2 + auricular electrode + conductive gel) 25 Hz stimulation will be applied, intensity escalated up to 15 mA or below if tingling sensation.

tVNS will be performed 1 hour daily for 1 month and we will assess EHOA symptoms (pain and function) at 1 month (end of the study)

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Symptomatic HOA (1990 American College of Rheumatology criteria)
* EHOA according to hand radiographs with ≥1 erosive digital joints of proximal or distal interphalangeal joint (phases "E" or "R" of Verbruggen-Veys score)
* Visual Analogic Scale (VAS) for hand pain ≥ 40/100 at inclusion

  -≥1 interphalangeal joints symptomatic ≥ 3 months despite analgesics or non-steroidal anti-inflammatory drugs (NSAIDs) (or contraindicated)
* ≥1 symptomatic interphalangeal joint with clinical palpable synovitis at inclusion
* Informed written consent

Exclusion Criteria:

* Isolated thumb-base OA (ie, rhizarthrosis)
* Hand osteoarthritis secondary to other known causes (eg gout, psoriatic arthritis)
* Psoriasis
* Current skin disease of the ear
* Ear canal not adapted to apply the auricular electrode
* History of severe cardiac disease (coronary artery disease, rhythm disturbance, heart failure, valvulopathy)
* Conduction or rhythm disturbances on electrocardiogram
* Symptomatic orthostatic hypotension or vasovagal syncope history
* History of vagotomy
* Pregnancy
* Fibromyalgia
* Use of other electrically active medical devices (eg pacemaker)
* Documented sleep apnea
* Use of corticosteroid (oral, intramuscular, intra-articular or intravenous), immunosuppressive agents, hyaluronic acid injection in interphalangeal joint within the last 3 months
* Hand surgery planned during the study period
* Pregnancy or breastfeeding if applicable
* Oral NSAIDs consumption during the last 48 hours before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Measure of Pain | 1 month
  Self-reported hand pain in the previous 48h measured on a 100 mm visual analogic scale (VAS).
  Scoring system:
  0= No pain 5= Moderate pain 10= Worst pain

SECONDARY OUTCOMES:
Function | 1 month
  questionnaire Functional Index for Hand OsteoArthritis (FIHOA): scale minimum 0 , and maximum 30.
  Scoring system of the FIHOA:
  0 = possible without difficulty
  1. = possible with slight difficulty
  2. = possible with important difficulty
  3. = impossible
Side effect | 1 month
  Safety : report of side effects during the study period
Mean time of daily use and cumulative time of use from the device's tracker | 1 month
  Observance : Mean time of daily use and cumulative time of use during the 30 days before the 1 month visit collected from the device's tracker
Dose of daily consumption of paracetamol | 1 month
  Measure of Pain by daily consumption of paracetamol

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie Sellam, MD PhD PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Rheumatology department Saint-Antoine Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No